CLINICAL TRIAL: NCT00232557
Title: Effectiveness of a Telecommunications System in Asthma Management
Brief Title: Telecommunications System in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 01-054
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
Keywords: Asthma; Disease Management; Telecommunications; Health Services; Quality of Life; Patient Compliance
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TLC-Asthma (Experimental): Telephone-based home education and asthma monitoring
  Interventions: Device: TLC-Asthma
- TLC-health education (Active Comparator): Telephone-based home education
  Interventions: Device: TLC-health education

INTERVENTIONS:
Device: TLC-Asthma — Telephone-linked communication (TLC) designed to improve asthma self-management by enhancing compliance with preventive medication regimens
  Arms: TLC-Asthma
Device: TLC-health education — A telephone-linked communication system (TLC) to provide general health education.
  Arms: TLC-health education

SUMMARY:
This project is investigating whether application of a telecommunications system to the care of adult patients with asthma will improve self-management by enhancing compliance with preventive medication regimens and fostering the use of peak-flow-based action plans.

DETAILED DESCRIPTION:
Background/Rationale:

Asthma is one of the most common chronic diseases of adults, affecting 6% of the U.S. adult population and accounting for substantial morbidity and mortality. Despite the availability of effective therapy for asthma, morbidity and mortality have increased over the last several decades. Asthma specialty care, case management, and patient education are means for improving the quality of asthma care and patient outcomes, but cost and inconvenience limit the degree to which these are used in asthma care nationally. The principal aim of this study is to evaluate the impact of an inexpensive telephone-based home education and disease monitoring system on asthma medication adherence and clinical outcomes in adult patients with asthma.

Objective(s):

We hypothesize that application of TLC to the care of adult patients with asthma will improve self-management by enhancing compliance with preventive medication regimens and fostering the use of peak flow-based action plans. This, in turn, will improve asthma control, thus reducing acute health care utilization and improving quality of life (QOL).

Methods:

A randomized controlled trial will be conducted with adult asthma patients identified from the VA Boston Healthcare System comprised of the Boston, West Roxbury, and Brockton VA Medical Centers and their associated satellite clinics. Patients will be randomized to either the TLC-Asthma group or an attention placebo control group. Outcome measurements will include medication adherence, QOL, utilization of urgent care services, oral corticosteroid use.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma
* Receiving treatment with one or more daily controller (i.e., preventive) medications
* Age = 18 years
* Less than 30 pack years of cigarette smoking
* FEVi greater than 50% of predicted
* FEVi bronchodilator response of at least 12%
* Ability to use a telephone without assistance

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TLC-Asthma: A telephone-linked communication (TLC) system to improve asthma self-management by enhancing compliance with preventive medication regimens
- TLC-health Education: A TLC system for providing general health education
Period: Overall Study
Arm/Group | TLC-Asthma | TLC-health Education
Started | 71 | 65
Completed | 68 | 60
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Population: Subject with baseline examination
Groups:
- Total: Total of all reporting groups
Arm/Group | TLC-Asthma | TLC-health Education | Total
Number analyzed (Participants) | 71 | 65 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (13.9) | 62.8 (14.3) | 61.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Participants With Unscheduled Asthma-related Visits
Description: Number of participants found to have any unscheduled office visits, emergency room visits, or hospitalizations that are related to asthma during one year.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | TLC-Asthma | TLC-health Education
Number analyzed (Participants) | 71 | 65
participants | 29 | 26

2. Secondary Outcome: Participants With Oral Corticosteroid Use
Description: Number of participants found to have any use of oral corticosteroids related to asthma during one year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | TLC-Asthma | TLC-health Education
Number analyzed (Participants) | 71 | 65
participants | 14 | 19

ADVERSE EVENTS:
Groups:
- Arm 1: A telephone-linked communication (TLC) system to improve asthma self-management by enhancing compliance with preventive medication regimens
- Arm 2: A TLC system for providing general health education
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/65
Other Adverse Events (participants affected / at risk) | 0/71 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes